CLINICAL TRIAL: NCT01350531
Title: Interventionist Procedures for Adherence to Weight Loss Recommendations in Black Adolescents, Phase Two
Brief Title: Interventionist Procedures for Adherence to Weight Loss Recommendations in Black Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Sylvie Naar-King, Ph.D., Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1U01HL097889 (NIH)
Record Dates: First submitted 2011-04-21; First posted 2011-05-09 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-01

CONDITIONS: Obesity
Keywords: Obesity; African American adolescents; Motivation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Skills training (Experimental)
  Interventions: Behavioral: Skills training
- Contingency Management (Experimental)
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Skills training — This component includes skills most proximal to adhering to the eating and weight loss plan (e.g., calorie counting, making healthy food choices, measuring food portions, scheduling snacks and meals, meal planning, completing food logs daily, following an exercise plan).
  Arms: Skills training
Behavioral: Contingency Management — Contingency management uses behavioral principles to counteract the reinforcing mechanisms of food and inactivity.
  Arms: Contingency Management

SUMMARY:
To date, attempts to construct effective weight loss interventions for African American adolescents with obesity (AAAO) have largely failed. While effective weight loss strategies and skills have been identified, lifestyle changes require youth and their families to learn new dietary and exercise behavior with repeated skills practice in natural ecology of the family. A major barrier is motivation of both parents and adolescents to engage in treatment and to adhere to behavior change recommendations. Advances in the science of increasing human motivation (both intrinsic and extrinsic) that could inform intervention development for minority youth with obesity have been insufficiently applied to date to the process of intervention development. The study brings together a multidisciplinary research group comprised of obesity intervention researchers with extensive experience in adolescent health behavior change research, basic behavioral scientists with experience in motivation and learning research and communication scientists with experience in provider-family interactions within urban populations. Basic science obesity researchers will inform intervention development by contributing a strong background in the physiological correlates of obesity. Finally experts in the area of community interventions for African American adolescents will contribute to the effective transport of these interventions to real-world settings. The overarching aims of the study are: To refine intervention protocols from our preliminary studies that maximize adolescent and parent skills, informed by learning theory, through the use of home and community-based interventions in which in-vivo opportunities are used to promote practice in making changes in dietary, exercise and sedentary behaviors in AAAO and their families (PHASE I); To develop intervention protocols that utilize findings from basic science regarding intrinsic and extrinsic motivation to maximize adolescent and family adherence to recommendations for obesity-related behavior change in AAAO and their families (PHASE I); To develop an adaptive intervention using a sequential multiple randomized assignment trial (SMART design) (PHASE II); To refine the intervention including qualitative analysis of interviews from participant families and to develop further community participation in preparation for a confirmatory randomized clinical trial (PHASE III).

There are two proposed hypotheses for this study:

1. Families initially receiving home/community delivery of Motivational Interviewing (MI)/skills training will show greater weight loss over the course of the study than families receiving initial office-based delivery of MI/skills training.
2. Non-responders receiving home/community delivery of MI/skills training with Contingency Management (CM) will show greater weight loss than non-responders receiving MI/skills training alone.

ELIGIBILITY:
Inclusion Criteria:

1. African American adolescents age range from 12 years to 16 years and 11 months with obesity (BMI>=95th percentile or BMI>30).
2. Adolescents may have primary obesity or obesity in combination with other medical co-morbidities.
3. Youth with mild mental retardation may be included if they are capable of reading and understanding the study measures.

Exclusion Criteria:

1. Obesity secondary to medication use for another disorder;
2. Obesity in a youth with medical condition that prevents their participation in normal exercise;
3. African American adolescent with obesity (AAAO) with thought disorders;
4. AAAO with serious cognitive impairments;
5. AAAO who are pregnant or have a medical condition where weight loss is contraindicated;
6. AAAO who do not live with their primary caregiver.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2009-09; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in weight-related outcomes at 6 months and 9 months | 6 months, 9 months
  We will be measuring participants' height, weight and percentage of body fat (Bioelectrical impedance analysis).

SECONDARY OUTCOMES:
Change from Baseline in Adherence to Weight Loss Recommendations at 6 months and 9 months. | 6 months, 9 months
  Objective measures of cardiovascular fitness will be used in addition to the BLOCK Kids Food Frequency Questionnaire, and the Frequency of Fast Food Use Questionnaire.
Change in Physiological Functioning from month 1 to 7 months | 1 month, 7 months
  Blood samples will be obtained after a 10-12 hour fast for measurement of plasma glucose, insulin, total cholesterol, high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), and triglyceride levels.
Change from Baseline in Motivation at 6 months and 9 months | 6 months, 9 months
  The Importance Ruler measure assesses how important different behaviors are to teens with regard to their weight loss. An analogous measure will be used to measure the importance of different behaviors in caregivers, as well.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Naar-King, Ph.D., Principal Investigator — Wayne State University; K-L Cathy Jen, Ph.D., Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Background] Albrecht TL, Ruckdeschel JC, Ray FL 3rd, Pethe BJ, Riddle DL, Strohm J, Penner LA, Coovert MD, Quinn G, Blanchard CG. A portable, unobtrusive device for videorecording clinical interactions. Behav Res Methods. 2005 Feb;37(1):165-9. doi: 10.3758/bf03206411. PMID 16097357
- [Background] Type 2 diabetes in children and adolescents. American Diabetes Association. Diabetes Care. 2000 Mar;23(3):381-9. doi: 10.2337/diacare.23.3.381. No abstract available. PMID 10868870
- [Background] Barlow SE; Expert Committee. Expert committee recommendations regarding the prevention, assessment, and treatment of child and adolescent overweight and obesity: summary report. Pediatrics. 2007 Dec;120 Suppl 4:S164-92. doi: 10.1542/peds.2007-2329C. PMID 18055651
- [Background] Barlow SE, Dietz WH. Obesity evaluation and treatment: Expert Committee recommendations. The Maternal and Child Health Bureau, Health Resources and Services Administration and the Department of Health and Human Services. Pediatrics. 1998 Sep;102(3):E29. doi: 10.1542/peds.102.3.e29. PMID 9724677
- [Background] Berwick DM. Disseminating innovations in health care. JAMA. 2003 Apr 16;289(15):1969-75. doi: 10.1001/jama.289.15.1969. PMID 12697800
- [Background] Block G, Woods M, Potosky A, Clifford C. Validation of a self-administered diet history questionnaire using multiple diet records. J Clin Epidemiol. 1990;43(12):1327-35. doi: 10.1016/0895-4356(90)90099-b. PMID 2254769
- [Derived] Naar S, Chapman J, Cunningham PB, Ellis D, MacDonell K, Todd L. Development of the Motivational Interviewing Coach Rating Scale (MI-CRS) for health equity implementation contexts. Health Psychol. 2021 Jul;40(7):439-449. doi: 10.1037/hea0001064. PMID 34435795
- [Derived] Lee MS, Carcone AI, Ko L, Kulik N, Ellis DA, Naar S. Managing Outliers in Adolescent Food Frequency Questionnaire Data. J Nutr Educ Behav. 2021 Jan;53(1):28-35. doi: 10.1016/j.jneb.2020.08.002. Epub 2020 Oct 1. PMID 33012663
- [Derived] Jacques-Tiura AJ, Ellis DA, Idalski Carcone A, Naar S, Brogan Hartlieb K, Towner EK, N Templin T, Jen KC. African-American Adolescents' Weight Loss Skills Utilization: Effects on Weight Change in a Sequential Multiple Assignment Randomized Trial. J Adolesc Health. 2019 Mar;64(3):355-361. doi: 10.1016/j.jadohealth.2018.09.003. Epub 2018 Nov 2. PMID 30392864
- [Derived] Hartlieb KB, Jacques-Tiura AJ, Naar-King S, Ellis DA, Jen KL, Marshall S. Recruitment strategies and the retention of obese urban racial/ethnic minority adolescents in clinical trials: the FIT families project, Michigan, 2010-2014. Prev Chronic Dis. 2015 Feb 19;12:E22. doi: 10.5888/pcd12.140409. PMID 25695260